CLINICAL TRIAL: NCT05804045
Title: A Phase 3, Randomized, Double-blind, Placebo-Controlled, Multicenter Study of ABSK021 to Assess the Efficacy and Safety in Patients With Tenosynovial Giant Cell Tumor
Brief Title: Study of Pimicotinib (ABSK021) for Tenosynovial Giant Cell Tumor (MANEUVER)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABSK021-301
Record Dates: First submitted 2023-03-13; First posted 2023-04-07 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Tenosynovial Giant Cell Tumor; Pigmented Villonodular Synovitis; Giant Cell Tumor of Tendon Sheath
MeSH Terms: conditions — Giant Cell Tumor of Tendon Sheath; Synovitis, Pigmented Villonodular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1/Part 2/Part 3- Pimicotinib(ABSK021)/ Pimicotinib(ABSK021) (Experimental): Participants receive the blinded treatment of ABSK021 for 24 weeks in Part 1 and continue on the open-label Pimicotinib(ABSK021) in Part 2 and Part 3.
  Interventions: Drug: Pimicotinib(ABSK021)
- Part 1- Placebo/ Pimicotinib(ABSK021) (Placebo Comparator): Participants receive the blinded treatment of matching placebo for 24 weeks in Part 1 and have option to receive the open-label Pimicotinib(ABSK021) in Part 2.
  Interventions: Drug: Pimicotinib(ABSK021); Drug: Placebo

INTERVENTIONS:
Drug: Pimicotinib(ABSK021) — capsule
Drug: Placebo — capsule
  Arms: Part 1- Placebo/ Pimicotinib(ABSK021)

SUMMARY:
The goal of this clinical trial is to assess the efficacy and safety of Pimicotinib (ABSK021) in patients with Tenosynovial Giant Cell Tumor (TGCT). The main questions it aims to answer are:

* Whether the Pimicotinib(ABSK021) works well in patients with TGCT.
* Whether the Pimicotinib(ABSK021) is safe in patients with TGCT.

Participants will be asked to complete the study procedures:

* Receive the administration of Pimicotinib(ABSK021) or placebo (a placebo is a look-alike substance that contains no active drug) about 24 weeks in study part 1.
* Receive the administration of Pimicotinib(ABSK021) about 24 weeks in study part 2.
* Receive the administration of Pimicotinib(ABSK021) till study end in study part 3.
* Complete the study procedures speficied in the protocol, which is guided by researchers.

DETAILED DESCRIPTION:
This study consists of part 1 and part 2. Part 1 is a double-blind phase, eligible patients will be randomized to Pimicotinib(ABSK021) treatment group or matching placebo group and will receive Pimicotinib(ABSK021) or matching placebo until completion of Part 1.

Part 2 is an open-label treatment phase, and all patients entering this phase will receive open-label Pimicotinib(ABSK021) until completion of 24 weeks of dosing or withdrawal from the study.

Part 3 is an open-label extension treatment phase, and patients who completed the part 2 and continuted to be eligible, will go to the Part 3. Patients will receive the open-label Pimicotinib(ABSK021) until all patients withdraw from the study, or the sponsor decides to terminate the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients should understand the study procedures and sign the informed consent form prior to screening.
* Age ≥ 18 years.
* A histologically confirmed TGCT with unresectable.
* Measurable disease as defined by RECIST 1.1, and with at least one lesion of ≥ 2 cm.
* Stable prescription of analgesic regimen for patients with an analgesic need.
* Participants should complete stiffness and pain scales during the screening period, and symptomatic disease because of active TGCT should meet minimum requirements as outlined in study protocol.
* ECOG PS (Eastern Cooperative Oncology Group Performance Status) of 0 or 1.
* Adequate organ function and bone marrow function.

Exclusion Criteria:

* Known allergy or hypersensitivity to any components of the investigational drug product.
* Previous treatment with highly selective inhibitors targeting CSF-1/CSF-1R. Previous therapy with imatinib and nilotinib is allowed.
* Known additional malignancy that required active treatment and may affect the patient's participation in the study or affect the outcome of the study as assessed by the Investigator.
* Known metastatic TGCT.
* Significant concomitant arthropathy in the affected joint, serious disease, uncontrolled infection.
* Known MRI contraindications.
* Has factors that significantly affected the absorption of oral drug.
* Major surgery or previous anti-tumor therapy for TGCT within 4 weeks prior to randomization.
* Concomitant use of strong CYP inhibitors or inducers as outlined in study protocol.
* Impaired cardiac function or clinically significant cardiac disease.
* Known active human immunodeficiency virus, active hepatitis B, active hepatitis C, or known active tuberculosis.
* Known active liver or biliary disease, or other diseases that may lead to abnormal liver function test results during the study.
* Pregnant or lactating women.
* Childbearing potential males or non-surgically sterilized female patients must agree to use effective methods of contraception during the study.
* Any other clinically significant comorbidities, which in the judgment of the Investigator, could compromise compliance with the protocol, interfere with the interpretation of study results, or predispose the patient to safety risks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Baseline to Week 25
  Assessed by central read using Response Evaluation Criteria in Solid Tumors (RECIST) (Version 1.1)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per Tumor Volume Score (TVS) | Baseline to Week 25
  Assessed by central read using Tumor Volume Score (TVS). TVS is a semi-quantitative MRI scoring system that describes tumor mass and is based on 10% increments of the estimated volume of the maximally distended synovial cavity or tendon sheath involved. A tumor that is equal in volume to that of a maximally distended synovial cavity or tendon sheath was scored 10; a score of 0 indicated no evidence of tumor.
Range of Motion (ROM) | Baseline to Week 25
  Mean change from baseline in ROM of the affected joint
Worst Stiffness | Baseline to Week 25
  Mean change from baseline in the Worst Stiffness Numeric Rating Scale (NRS) score at Week 25. The Worst Stiffness Numeric Rating Scale (NRS) was a 1-item, self-administered questionnaire assessing the "worst" stiffness in the last 24 hours. The NRS for this item ranged from 0 (no stiffness) to 10 (stiffness as bad as you can imagine). Higher scores mean a worse outcomes.
Worst Pain | Baseline to Week 25
  Mean change from baseline in the Worst Pain Numeric Rating Scale (NRS) score at Week 25. The Worst Pain Numeric Rating Scale Score (NRS) was a 1-item, self-administered questionnaire assessing the "worst" pain in the last 24 hours. The NRS for this item ranged from 0 (no pain) to 10 (pain as bad as you can imagine). Higher scores mean a worse outcomes.
Physical Function | Baseline to Week 25
  Mean change from baseline in the Patient-reported Outcomes Measurement Information System (PROMIS) Physical Function score at Week 25. The Patient-reported Outcomes Measurement Information System (PROMIS) physical function scale was used to assess physical function of the upper and lower limbs. The scale ranged from 1 defined as 'unable to do' or 'cannot do' to 5 defined as 'without any difficulty' or 'not at all', where higher scores represent better outcomes.
Quality of life (QoL) | Baseline to Week 25
  Mean change from baseline in EuroQol visual analogue scale (VAS) score at Week 25. The EuroQol visual analogue scale (VAS) is a Visual Analogue Scale on which the patient rates their current health, with 0 representing the "worst health you can imagine" and 100 representing the "best health you can imagine". Higher scores mean a better outcomes.
Duration of Response (DOR) | The time (months) from the first documentation of objective response to the first documentation of radiographic disease progression (PD) or death due to any cause, whichever occurs first, assessed up to 24 months.
  Duration of Response as measured by RECIST Version 1.1 and Tumor Volume Score (TVS)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (8):
  - Precision NextGen Oncology, Beverly Hills, California
  - Duke University Medical Center, Durham, California
  - Henry Ford Health System, Detroit, Michigan
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Canada (2):
  - McGill University Health Center, Montreal
  - Princess Margaret Cancer Center, Toronto
- China (23):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The Central Hospital of Enshi Tujia and Miao Autonomous Prefecture, Enshi, Hubei
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Drum Tower hospital, Nanjing, Jiangsu
  - Liaoning Cancer Hospital&Institute, Shenyang, Liaoning
  - Weifang People's Hospital, Weifang, Shandong
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Xi'an Honghui Hospital, Xi’an, Shanxi
  - West China Hospital Sichuan University, Chengdu, Wuhan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Beijing Jishuitan Hospital, Beijing
- Italy (3):
  - IRCCS Istituto Ortopedico Rizzoli, Bologna
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Ospedale di Prato, Prato
- Leiden University Medical Center, Leiden, Netherlands
- Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw, Poland
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Fundacion Jimenez Diaz, Madrid

REFERENCES:
- [Derived] Niu X, Ravi V, Shan B, Guo Q, Shi H, Zou Q, Gelderblom H. MANEUVER: A Phase III study of pimicotinib to assess efficacy and safety in tenosynovial giant cell tumor patients. Future Oncol. 2024 Sep 17:1-8. doi: 10.1080/14796694.2024.2396227. Online ahead of print. PMID 39287124